CLINICAL TRIAL: NCT03157076
Title: BIO|CREATE Pilot Study
Brief Title: Pilot Study to Investigate the Creation of Physiological Rhythm by Closed Loop Stimulation in hEart Failure pAtients With chronoTropic incompEtence
Acronym: BIO|CREATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR019
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure; CPX
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Intervention Model Description: Patients are randomized in two different pacing modes (CLS versus intrinsic rhythm) after one month after enrollment. The cross-over takes place after one month after the randomization.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pacing mode with CLS (Active Comparator)
  Interventions: Device: Cardiac Resynchronization therapy device with Closed Loop Stimulation (CLS)
- Intrinsic mode (Active Comparator)
  Interventions: Device: Cardiac Resynchronization therapy device with Closed Loop Stimulation (CLS)

INTERVENTIONS:
Device: Cardiac Resynchronization therapy device with Closed Loop Stimulation (CLS) — The feature CLS will be programmed ON or Off according to a randomization list after one month after baseline visit. One month later the alternate will be programmed.
  Other Names: Cardiac Resynchronization therapy device without Closed Loop Stimulation (CLS)

SUMMARY:
The study assesses the effect of Closed Loop Stimulation (CLS) on the ventilatory efficiency slope and estimates the patient responder rate to CLS in patients with severe chronotropic incompetence treated with a cardiac resynchronization therapy (CRT) device.

DETAILED DESCRIPTION:
In patients with pharmacological refractory heart failure (HF), systolic dysfunction, and cardiac dyssynchrony, the cardiac resynchronization therapy (CRT) reduces the risk of death, and improves symptoms and quality of life.

A considerable portion (80%) of patients with a CRT indication has a chronotropic incompetence (CI). CI usually induces a stress intolerance which negatively affects the quality of life. In addition of being a marker of diminished exercise capacity, severe CI (sCI) may be an independent predictor of mortality.

The sensor-based rate adaption provided by the implanted CRT device delivers a possible therapeutic approach for the CI.

Usually, rate adaption is achieved by an accelerometer. The previous studies in terms of effectiveness of rate adaption in CRT patients with CI showed inconsistent results.

In addition to an accelerometer to deliver the rate adaption BIOTRONIK provides closed loop stimulation (CLS) as unique feature in a CRT device. CLS determines the appropriate heart rate based on intra-cardiac impedance measurements. These measurements reflect changes of the cardiac contraction dynamics in reaction to information coming from the autonomic nervous system. CLS takes the information on the contraction dynamics and translates it into an adequate heart rate adaptation, thus delivering physiologically appropriate therapy.

ELIGIBILITY:
Inclusion Criteria:

* CRT class I indication at time of implantation, according to current guidelines
* Implantation of CRT-device including CLS > 6 months prior to enrollment
* Stable heart failure status for at least 1 month
* Optimal cardiovascular drug treatment according to current guidelines
* NYHA class II or III
* Patient is able to comply with the protocol
* Patient provided written informed consent
* Stable location of residence

Exclusion Criteria:

* Planned cardiovascular intervention within the next 3 months
* Admission for decompensated heart failure or acute coronary syndrome in the preceding 3 months
* Ongoing symptoms of myocardial ischemia
* Known persistent, long-standing persistent or permanent atrial fibrillation
* COPD with GOLD ≥ 3
* Planned absence of residence for more than one week during study period
* Pregnant or breast-feeding women
* Participation in another interventional clinical investigation
* Age < 18 years
* Placed in an institution due to official decree or judicial order
* Dependent from the sponsor, the clinical site or the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Ventilatory efficiency slope | 2 months
  The slope of VE/VCO2 describes the ventilatory efficiency during effort, showing the amount of air that must be ventilated to eliminate 1 litre of CO2.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Roser, Dr., Principal Investigator — Charité Universitätsklinikum - Campus Benjamin Franklin
Locations (1):
- Charité Universitätsklinikum - Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No